CLINICAL TRIAL: NCT04538248
Title: Efficiency of Combined Rehabilitation Programs Including Resistance and Endurance Exercises on Functional Capacities, Quality of Life and Daily Level of Activities in Hemodialysis Patients: a Comparative Study of Current Practices.
Brief Title: Efficiency of Combined Rehabilitation Programs Including Resistance and Endurance Exercises on Functional Capacities, Quality of Life and Daily Level of Activities in Hemodialysis Patients
Acronym: DIALEX
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0403
Record Dates: First submitted 2020-09-02; First posted 2020-09-04 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Chronic Kidney Diseases; Hemodialysis; Physical Rehabilitation
Keywords: Perdialytic exercise; Combined rehabilitation; Functional abilities; Interference effect
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Continuous: Continuous
  Interventions: Other: Combined rehabilitation during hemodialysis
- Discontinuous: Discontinuous
  Interventions: Other: Combined rehabilitation during hemodialysis

INTERVENTIONS:
Other: Combined rehabilitation during hemodialysis — Combined rehabilitation during hemodialysis

SUMMARY:
Hemodialysis patients display among the lowest level of daily activities and decline of functional abilities is highly correlated with mortality. Perdialytic exercise during hemodialysis procedure is now part of the patients' routine care and appears to be a solution to struggle against the functional skills decrease. Our team was able to demonstrate that beyond muscle mass, muscle strength and physical activity were essential determinants of morbidity and mortality of dialysis patients. The AIDER Santé medical team has set up an assessment of physical activities and muscle strength in the Montpellier and Nimes centers. In order to rehabilitate muscle strength and endurance, perdialytic exercise may be prescribed. Its effectiveness can be appreciated by measuring the SPPB score (Short Physical Performance Battery). Recent studies established that combined training including resistance and endurance exercises was the most effective to improve functional performance. In AIDER Santé dialysis centers, the two mainly used exercise approaches are distinguished by the time distribution of the two types of exercise: the first plans to practice both types of exercise at each session (continuous program), the second plans to alternate a week of resistance exercise with a week of endurance exercise (discontinuous program). It is established that the rehabilitation of the hemodialysis patient must include both resistance and endurance exercises, but the combination of these exercises during the same session is potentially at the origin of an interference phenomenon, limiting neuromuscular adaptations specific to each effort. Therefore, the main hypothesis of the project is that the temporal separation of resistance and endurance exercises in a discontinuous program could optimize the functional gains of combined rehabilitation and therefore be more effective than a continuous program generating a phenomenon of interference.

ELIGIBILITY:
Inclusion criteria:

* Hemodialysis started since at least 3 months
* Medical prescription of perdialytic combined exercise
* Age < 85
* Life expectancy > 6 months

Exclusion criteria:

* Ischemic and valvular cardiopathies
* Lower-extremity arterial disease (stade III and IV)
* Knee or hip amputation/prothesis
* Severe respiratory disease
* BMI > 35
* Pacemaker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients of Montpellier AIDER Santé dialysis center
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Short Physical | Week 0, week 17
  Short Physical Performance Battery Score

SECONDARY OUTCOMES:
Knee extension force | 1 day
  Knee extension force

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Principal Investigator — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No